CLINICAL TRIAL: NCT00092716
Title: A Multicenter, Double-Blind, Randomized, Parallel Group, 28-Week Study to Evaluate the Efficacy and Safety of Ezetimibe and Simvastatin Co-administration Versus Atorvastatin in Patients With Hypercholesteremia
Brief Title: Comparing an Investigational Medication Versus an Approved Medication in Reducing Cholesterol Levels (0653-025)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-025; 2004_047
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Duration of Therapy

INTERVENTIONS:
Drug: MK0653, ezetimibe / Duration of Treatment: 28 weeks
Drug: Comparator: atorvastatin / Duration of Treatment: 28 weeks

SUMMARY:
The purpose of this study is to determine whether an investigational medication will be more effective than an approved medication in reducing cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Elevated cholesterol levels

Exclusion Criteria:

* Liver disease
* Unstable medical conditions

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2002-05; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect on the reduction in low density lipoprotein cholesterol (LDL-C) after the initial 6-week treatment period.

SECONDARY OUTCOMES:
Assess safety/tolerability and evaluate effect on HDL-C & on reduction of LDL-C
Evaluate % of pts who attain their NCEP-ATP III goal for LDL-C @ each dose level

REFERENCES:
- [Background] Ballantyne CM, Blazing MA, King TR, Brady WE, Palmisano J. Efficacy and safety of ezetimibe co-administered with simvastatin compared with atorvastatin in adults with hypercholesterolemia. Am J Cardiol. 2004 Jun 15;93(12):1487-94. doi: 10.1016/j.amjcard.2004.02.060. PMID 15194018
- [Background] McKenney J, Ballantyne CM, Feldman TA, Brady WE, Shah A, Davies MJ, Palmisano J, Mitchel YB. LDL-C goal attainment with ezetimibe plus simvastatin coadministration vs atorvastatin or simvastatin monotherapy in patients at high risk of CHD. MedGenMed. 2005 Jul 14;7(3):3. PMID 16369229
- [Background] Catapano A, Brady WE, King TR, Palmisano J. Lipid altering-efficacy of ezetimibe co-administered with simvastatin compared with rosuvastatin: a meta-analysis of pooled data from 14 clinical trials. Curr Med Res Opin. 2005 Jul;21(7):1123-30. doi: 10.1185/030079905X50642. PMID 16004682